CLINICAL TRIAL: NCT03692052
Title: A Phase 2, Open-label, Multicenter Study to Determine the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of AG-348 in Adult Subjects With Non-transfusion-dependent Thalassemia
Brief Title: A Study to Determine the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of AG-348 in Adult Participants With Non-transfusion-dependent Thalassemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-010; 2018-002217-35 (EudraCT Number)
Record Dates: First submitted 2018-09-10; First posted 2018-10-02 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG-348 (Experimental): Participants with alpha or beta thalassemia received AG-348 50 mg twice daily (BID), orally up to Week 6. Following Week 6, depending on the participants' safety and hemoglobin (Hb) concentrations, they could undergo one potential dose-level increase from 50 to 100 mg BID. After completion of the Core Period of 24 weeks, participants were eligible to continue to receive AG-348 in the Extension Period which is up to 10 years.
  Interventions: Drug: AG-348

INTERVENTIONS:
Drug: AG-348 — AG-348 tablet orally BID
  Other Names: Mitapivat

SUMMARY:
Study AG348-C-010 is a multicenter study to evaluate the efficacy, safety, pharmacokinetics, and pharmacodynamics of treatment with AG-348 in adult participants with non-transfusion-dependent thalassemia (NTDT). This study includes a core period (up to 24 weeks) followed by an extension period (up to 10 years) for eligible participants. 20 participants with NTDT were enrolled. The initial dose of AG-348 was 50 milligrams (mg) twice daily (BID) with one potential dose-level increase to 100 mg BID at the Week 6 visit based on the participant's safety and hemoglobin (Hb) concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent;
* Known medical history of thalassemia, including β-thalassemia intermedia, Hb E β-thalassemia, α-thalassemia (Hb H disease), or β-thalassemia with mutations of 1 or more α genes;
* Documented clinical laboratory confirmation of thalassemia by Hb electrophoresis/high-performance liquid chromatography (HPLC) or deoxyribonucleic acid (DNA) analysis, either from medical records or during the screening period;
* Hb concentration ≤10.0 grams per deciliter (g/dL), regardless of sex, based on an average of at least 2 Hb measurements (separated by a minimum of 7 days) during the screening period;
* Considered non-transfusion-dependent, defined as having no more than 5 units of red blood cells (RBCs) transfused during the 24-week period up to the first day of study drug and no RBC transfusions in the 8 weeks prior to the first day of study drug;
* Adequate organ function;
* For women of reproductive potential: negative serum pregnancy test during the screening period and a negative serum or urine pregnancy test on Day 1;
* For women of reproductive potential as well as men with partners who are women of reproductive potential: be abstinent as part of their usual lifestyle, or agreement to use 2 forms of contraception, 1 of which must be considered highly effective, from the time of giving informed consent, during the study, and for 28 days following the last dose of study drug for women and 90 days following the last dose of study drug for men;
* Willingness to comply with all study procedures for the duration of the study;

Exclusion Criteria:

* Known history of diagnosis of Hb S or Hb C forms of thalassemia;
* Significant medical condition that confers an unacceptable risk to participating in the study, and/or could confound the interpretation of the study data;
* Splenectomy scheduled during the study treatment period or having undergone splenectomy within 12 months prior to signing informed consent;
* Currently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo;
* Exposure to any investigational drug, device, or procedure within 3 months prior to the first day of study drug;
* Prior exposure to sotatercept (ACE-011), luspatercept (ACE-536), ruxolitinib, or gene therapy;
* Prior bone marrow or stem cell transplant;
* Currently pregnant or breastfeeding;
* History of major surgery within 6 months of signing informed consent;
* Currently receiving medications that are strong inhibitors of cytochrome P450 (CYP)3A4, strong inducers of CYP3A4, strong inhibitors of P-glycoprotein (P-gp), or digoxin (a P-gp sensitive substrate medication) that have not been stopped for a duration of at least 5 days or a timeframe equivalent to 5 half-lives (whichever is longer) prior to the first day of study drug;
* Currently receiving chronic anticoagulant therapy, unless started and on a stable dose for at least 28 days prior to first day of study drug;
* Currently receiving anabolic steroids, including testosterone preparations, if initiated ≤28 days prior to the first day of study drug;
* Currently receiving hematopoietic stimulating agents (e.g., erythropoietins, granulocyte colony stimulating factors, thrombopoietins), if initiated ≤8 weeks prior to the first day of study drug;
* History of allergy to sulfonamides if characterized by acute hemolytic anemia, drug-induced liver injury, anaphylaxis, rash of erythema multiforme type or Stevens-Johnson syndrome, cholestatic hepatitis, or other serious clinical manifestations;
* History of allergy to AG-348 or its excipients (microcrystalline cellulose, croscarmellose sodium, sodium stearyl fumarate, and mannitol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2030-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (4):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Massachusetts General Hospital, Boston, Massachusetts
- University Health Network (Toronto General Hospital), Toronto, Ontario, Canada
- Imperial College Healthcare NHS Trust (Hammersmith Hospital), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuo KHM, Layton DM, Lal A, Al-Samkari H, Bhatia J, Kosinski PA, Tong B, Lynch M, Uhlig K, Vichinsky EP. Safety and efficacy of mitapivat, an oral pyruvate kinase activator, in adults with non-transfusion dependent alpha-thalassaemia or beta-thalassaemia: an open-label, multicentre, phase 2 study. Lancet. 2022 Aug 13;400(10351):493-501. doi: 10.1016/S0140-6736(22)01337-X. PMID 35964609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 4 investigative sites in the United States, Canada, and United Kingdom from 28 December 2018 to 30 September 2030. Results are reported for the primary and secondary outcome measures for the 24-week Core Period (data cut-off date: 20 August 2020). The Extension Period of this study is ongoing.
Pre-assignment Details: A total of 20 participants were enrolled in the Core Period of this study. The participants who completed the 24-week Core Period and achieved a hemoglobin (Hb) response or a delayed Hb response and had an acceptable safety profile were eligible to continue in the Extension Period.
Period: Core Period (Day 1 to Week 24)
Arm/Group | AG-348
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1
Period: Extension Period (Week 25 to 10 Years)
Arm/Group | AG-348
Started | 19
Completed | 0
Not Completed | 19
Not completed — Withdrawal of Consent | 1
Not completed — Physician Decision | 1
Not completed — Ongoing | 17

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study treatment.
Groups:
- AG-348: Participants with alpha or beta thalassemia received AG-348 50 mg BID, orally up to Week 6. Following Week 6, depending on the participants' safety and Hb concentrations, they could undergo one potential dose-level increase from 50 to 100 mg BID. After completion of the Core Period of 24 weeks, participants were eligible to continue to receive AG-348 in the Extension Period which is up to 10 years.
Arm/Group | AG-348
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Hemoglobin Response (HR)
Description: HR was defined as a ≥1.0 gram per deciliter (g/dL) increase in Hb concentration from Baseline at 1 or more assessments between Week 4 and Week 12 (inclusive). A participant's Baseline Hb concentration was defined as the average of all the participant's available Hb concentrations during the screening period up to the first dose of study drug.
Time Frame: Up to 12 weeks
Population: FAS included all participants who received at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 20
percentage of participants | 80.0 [59.90 to 92.86]
Statistical Analysis 1: Comparison: AG-348; Test type: Other; p < .0001, Clopper-Pearson Method; Significance of p-value associated with the test of H0:Hb response rate =0.3 vs H1:Hb response rate > 0.3

2. Secondary Outcome: Average Change From Baseline in Hb Concentrations From Week 12 to Week 24
Description: A participant's Baseline Hb concentration was defined as the average of all the participant's available Hb concentrations during the screening period up to the first dose of study drug.
Time Frame: Baseline, Week 12 to Week 24
Population: FAS included all participants who received at least 1 dose of study treatment. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | AG-348
Number analyzed (Participants) | 20
grams per liter (g/L)
  Baseline | 79.44 (13.690)
  Average Change from Baseline: Week 12 to 24: number analyzed (Participants) | 19
  Average Change from Baseline: Week 12 to 24 | 13.01 (6.283)

3. Secondary Outcome: Percentage of Participants Achieving a Sustained Hb Response (sHR)
Description: sHR was defined as achieving HR and achieving a ≥1.0 g/deciliter (dL) increase in Hb concentration at 2 or more evaluable Hb assessments out of the 4 scheduled assessments between the Week 12 visit and Week 24 visit.
Time Frame: Week 12 to Week 24
Population: FAS included all participants who received at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 20
percentage of participants | 65.0 [44.20 to 82.27]

4. Secondary Outcome: Percentage of Participants Achieving a Delayed Hb Response
Description: Delayed Hb response was defined as not achieving HR and achieving a ≥1.0 g/dL increase in Hb concentration at 1 or more Hb assessments after Week 12.
Time Frame: Week 12 to Week 24
Population: FAS included all participants who received at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 20
percentage of participants | 10.0 [1.81 to 28.26]

5. Secondary Outcome: Change From Baseline in Hb Concentration Over the Duration of the Extension Period
Time Frame: Baseline up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

6. Secondary Outcome: Time to First ≥1.0 g/dL Increase in Hb Concentration
Time Frame: Up to Week 24
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study treatment. Data is reported for the responders.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | AG-348
Number analyzed (Participants) | 16
weeks | 4.54 (3.204)

7. Secondary Outcome: Change From Baseline in Reticulocyte Count
Time Frame: Up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

8. Secondary Outcome: Change From Baseline in Bilirubin
Time Frame: Up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

9. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH)
Time Frame: Up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

10. Secondary Outcome: Change From Baseline in Haptoglobin
Time Frame: Up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

11. Secondary Outcome: Change From Baseline in Nucleated Red Blood Cells (NRBCs)
Time Frame: Up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

12. Secondary Outcome: Change From Baseline in Erythropoietin (EPO)
Time Frame: Up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

13. Secondary Outcome: Change From Baseline in Soluble Transferrin Receptor
Time Frame: Up to approximately 10.5 years
Reporting Status: Not Posted, anticipated posting 2031-09

14. Secondary Outcome: Drug Concentrations Over Time for AG-348
Time Frame: Predose (60 minutes) and 0.00 hour, 0.50 hour, 1 hour, 2 hours, 4 hours, and 8 hours postdose on Day 1 and Week 12
Population: The Pharmacokinetic (PK) Analysis Set included all participants who were enrolled and received a dose of study medication (AG-348), with at least one non-zero plasma concentration of AG-348 at Day 1 or Week 12 (or the Unscheduled Visit where intensive PK samples were assessed). Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | AG-348
Number analyzed (Participants) | 20
nanograms per milliliter (ng/mL)
  AG-348 50 mg: 0.00 Hour, Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: 0.00 Hour, Day 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable due to lower limit of quantitation.
  AG-348 50 mg: 0.50 Hour, Day 1: number analyzed (Participants) | 15
  AG-348 50 mg: 0.50 Hour, Day 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable due to lower limit of quantitation.
  AG-348 50 mg: 1 Hour, Day 1: number analyzed (Participants) | 17
  AG-348 50 mg: 1 Hour, Day 1 | 785.2 (64.6)
  AG-348 50 mg: 2 Hour, Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: 2 Hour, Day 1 | 694.5 (26.6)
  AG-348 50 mg: 4 Hour, Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: 4 Hour, Day 1 | 369.2 (29.4)
  AG-348 50 mg: 8 Hour, Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: 8 Hour, Day 1 | 128.9 (55.1)
  AG-348 100 mg: 0.00 Hour, Week 12: number analyzed (Participants) | 17
  AG-348 100 mg: 0.00 Hour, Week 12 | 39.39 (117.1)
  AG-348 100 mg: 0.50 Hour, Week 12: number analyzed (Participants) | 16
  AG-348 100 mg: 0.50 Hour, Week 12 | 1030 (137.7)
  AG-348 100 mg: 1 Hour, Week 12: number analyzed (Participants) | 12
  AG-348 100 mg: 1 Hour, Week 12 | 1442 (30.6)
  AG-348 100 mg: 2 Hour, Week 12: number analyzed (Participants) | 15
  AG-348 100 mg: 2 Hour, Week 12 | 740.1 (76.3)
  AG-348 100 mg: 4 Hour, Week 12: number analyzed (Participants) | 15
  AG-348 100 mg: 4 Hour, Week 12 | 302.8 (75.2)
  AG-348 100 mg: 8 Hour, Week 12: number analyzed (Participants) | 16
  AG-348 100 mg: 8 Hour, Week 12 | 77.35 (48.2)

15. Secondary Outcome: AUC0-8h: Area Under the Plasma Concentration-time Curve From Time 0 to 8 Hours of AG-348
Time Frame: Predose (60 minutes) and 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours postdose on Day 1 and Week 12
Population: The PK Analysis Set included all participants who were enrolled and received a dose of study medication (AG-348), with at least one non-zero plasma concentration of AG-348 at Day 1 or Week 12 (or the Unscheduled Visit where intensive PK samples were assessed). Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | AG-348
Number analyzed (Participants) | 20
nanograms*hour per milliliter (ng*h/mL)
  AG-348 50 mg: Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: Day 1 | 3083.3 (25.6)
  AG-348 100 mg: Week 12: number analyzed (Participants) | 15
  AG-348 100 mg: Week 12 | 3384.4 (65.7)

16. Secondary Outcome: AUC0-t: Area Under the Plasma Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration of AG-348
Time Frame: Predose (60 minutes) and 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours postdose on Day 1 and Week 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | AG-348
Number analyzed (Participants) | 20
ng*h/mL
  AG-348 50 mg: Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: Day 1 | 3083.5 (25.6)
  AG-348 100 mg: Week 12: number analyzed (Participants) | 15
  AG-348 100 mg: Week 12 | 3384.4 (65.7)

17. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration of AG-348
Time Frame: Predose (60 minutes) and 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours postdose on Day 1 and Week 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AG-348
Number analyzed (Participants) | 20
ng/mL
  AG-348 50 mg: Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: Day 1 | 968.9 (38.1)
  AG-348 100 mg: Week 12: number analyzed (Participants) | 16
  AG-348 100 mg: Week 12 | 1476 (93.5)

18. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Radioactivity Concentration (Cmax)
Time Frame: Predose (60 minutes) and 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours postdose on Day 1 and Week 12
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | AG-348
Number analyzed (Participants) | 20
hours
  AG-348 50 mg: Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: Day 1 | 1.07 [0.48 to 4.07]
  AG-348 100 mg: Week 12: number analyzed (Participants) | 16
  AG-348 100 mg: Week 12 | 0.53 [0.43 to 2.03]

19. Secondary Outcome: Tlast: Time of the Last Quantifiable Concentration of AG-348
Time Frame: Predose (60 minutes) and 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours postdose on Day 1 and Week 12
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | AG-348
Number analyzed (Participants) | 20
hours
  AG-348 50 mg: Day 1: number analyzed (Participants) | 19
  AG-348 50 mg: Day 1 | 7.60 [7.50 to 8.02]
  AG-348 100 mg: Week 12: number analyzed (Participants) | 15
  AG-348 100 mg: Week 12 | 7.55 [7.50 to 7.95]

20. Secondary Outcome: Ctrough: Observed Plasma Concentration at the End of a Dosing Interval of AG-348
Time Frame: Predose (60 minutes) and 30 minutes, 1 hour, 2 hours, 4 hours, and 8 hours postdose on Day 1 and Week 12
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | AG-348
Number analyzed (Participants) | 20
ng/mL
  AG-348 50 mg: Day 1: number analyzed (Participants) | 0
  AG-348 100 mg: Week 12: number analyzed (Participants) | 16
  AG-348 100 mg: Week 12 | 37.34 (117.7)

21. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), and TEAEs Leading to Study Drug Dose Reduction, Study Drug Interruption, and Study Drug Discontinuation
Description: An AE is any unfavorable and unintended sign, symptom, or disease, whether or not related to the investigational product. A TEAE was defined as any AE with onset post study drug treatment. An SAE was defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is medically important. AESIs are predefined AEs that required close monitoring and prompt reporting to the sponsor. AESIs included protocol-specified transaminase increase.
Time Frame: From signing the inform consent form up to data cut-off date: 20 August 2020 (Up to approximately 19 months)
Population: Safety Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | AG-348
Number analyzed (Participants) | 20
percentage of participants
  TEAEs | 85.0
  SAEs | 5.0
  AESIs | 5.0
  TEAEs Leading to Study Drug Dose Reduction | 15.0
  TEAEs Leading to Study Drug Interruption | 5.0
  TEAEs Leading to Study Drug Discontinuation | 5.0

ADVERSE EVENTS:
Time Frame: Up to completion of the Core Period data cut-off date: 20 August 2020 (Up to approximately 19 months)
Description: Safety Analysis Set included all participants who received at least 1 dose of study treatment.
Arm/Group | AG-348
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AG-348 (N=20)
Renal impairment (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AG-348 (N=20)
Initial insomnia (Psychiatric disorders) | 10
Anxiety (Psychiatric disorders) | 1
Middle insomnia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Terminal insomnia (Psychiatric disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 5
Carotid arteriosclerosis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 1
Fatigue (General disorders) | 4
Pain (General disorders) | 3
Chest discomfort (General disorders) | 2
Pyrexia (General disorders) | 2
Oedema peripheral (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Body tinea (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Suspected COVID-19 (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Ocular icterus (Hepatobiliary disorders) | 3
Aspartate aminotransferase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Fibrin D dimer increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/15 — Number at risk is based on the female population in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information obtained from the clinical study will be used towards the development of AG-348 and may be disclosed to regulatory authority(ies), other Investigators, corporate partners, or consultants as required.

DOCUMENTS (2):
  • Study Protocol (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT03692052/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03692052/SAP_001.pdf